CLINICAL TRIAL: NCT05282602
Title: Effects of Wii Fit Based Exercises and Proprioceptive Training on Balance and Fall Risk in Patients With Diabetic Neuropathy
Brief Title: Wii Fit Based Exercises and Proprioceptive Exercises in Diabetic Neuropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/22/0201 Maryam
Record Dates: First submitted 2022-02-20; First posted 2022-03-16 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Neuropathies
Keywords: Wii Fit; Proprioceptive; Fall; Balance; Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wii Fit Based Exercises (Experimental): Group A will receive Wii fit Based Exercises
  Interventions: Other: baseline physical therapy treatment along with Wii Fit based exercises
- Proprioceptive Training (Experimental): Group B will receive proprioceptive training
  Interventions: Other: Proprioceptive exercises

INTERVENTIONS:
Other: baseline physical therapy treatment along with Wii Fit based exercises — Group A performed Wii Fit based exercises for 6 weeks. Group A will be treated with Wii Fit based exercises (40 mins session, 3 days/week, Penguin slide, soccer heading, tilt table, tightrope walking)
  Arms: Wii Fit Based Exercises
Other: Proprioceptive exercises — Group B will be treated with Proprioceptive training (40 min session, 3 days/week, toe walking, heel walking, cross-body leg swings right and left sides, partial squat, ). In both groups pre and post-test measurements of Balance and Fall of risk will be assessed through Berg Balance scale, STAR excursion, Modified Fall Efficacy scale, and Timed Up and Go (TUG). Evaluation will be done before session start and at the end of 6th Week.
  Arms: Proprioceptive Training

SUMMARY:
This project is a Randomized clinical trial that will be conducted to check the effects of Wii Fit Based Exercises and Proprioceptive training on Balance and Fall Risk in patients with Diabetic Neuropathy, duration of study will be of 6months, convenient sampling will be used, subject following eligibility criteria from Riphah Rehabilitation Centre, Patients will be randomly allocated into two groups; Group A will be treated with Wii Fit based exercises (40 mins session, 3 days/week, Penguin slide, soccer heading, tilt table, tightrope walking) & Group B will be treated with Proprioceptive training (40 min session, 3 days/week, toe walking, heel walking, cross-body leg swings right and left sides, partial squat, ). In both groups pre and post-test measurements of Balance and Fall of risk will be assessed through Berg Balance scale, STAR excursion, Modified Fall Efficacy scale, and Timed Up and Go (TUG). Evaluation will be done before the session start and at the end of 6th Week.

DETAILED DESCRIPTION:
Diabetes mellitus is a disorder in which the body does not produce enough or respond normally to insulin, causing blood sugar (glucose) levels to be abnormally high. Diabetic neuropathy is a serious diabetes complication that may affect as many as 50% of people with diabetes. The nerve damage associated with diabetic peripheral neuropathy (DPN) may reduce the proprioceptive inputs that contribute to decreased balance and an increased risk of falling. Wii Fit Balance Board improves balance in older adults through training. Wii Fit balance board showed significant improvement in balance and decrease the risk of fall. Proprioceptive training is an intervention that targets the improvement of proprioceptive function in patients. The aim of the current study is to determine the effects of Wii Fit Based exercises and proprioception training on balance and fall of risk in patients with Diabetic Neuropathy

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age;
* Medical diagnoses of diabetes under regular medication control
* DN4 score ≥ 4
* Independent community ambulatory individuals;
* Intact cognition (Minimental State Examination score of >24

Exclusion Criteria:

* Other neurological diseases such as dementia, Parkinson's disease, spinal cord injury, or stroke;
* Severe visual impairment, musculoskeletal disorders, unhealed plantar ulceration, lower limb amputation, poor cardiopulmonary function, or other diseases affecting walking ability or any other disease due to which individuals were unable to walk without assistance
* Any other condition associated with a high risk of falling

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | 6th Week
  Determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling.
STAR Excursion test | 6th Week
  Functional screening tool to assess lower extremity dynamic stability and neuromuscular control
Modified Fall Efficacy scale | 6th Week
  Assess an individual's confidence in performing common activities of daily living without falling.5=fairly confident/fairly sure, and 10=completely confident/ completely sure. Scores can fall in between 0, 5, and 10. Interpretation: Higher scores reflect more confidence, less fear of falling. Lower scores reflect less confidence and more fear of falling
Timed Up and Go Test | 6th Week
  Assess a person's mobility and requires both static and dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, PhD, Study Chair — Riphah International University; Maryam Ikram, MSPT(NM)*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reeves ND, Orlando G, Brown SJ. Sensory-Motor Mechanisms Increasing Falls Risk in Diabetic Peripheral Neuropathy. Medicina (Kaunas). 2021 May 8;57(5):457. doi: 10.3390/medicina57050457. PMID 34066681
- [Background] Khan KS, Andersen H. The Impact of Diabetic Neuropathy on Activities of Daily Living, Postural Balance and Risk of Falls - A Systematic Review. J Diabetes Sci Technol. 2022 Mar;16(2):289-294. doi: 10.1177/1932296821997921. Epub 2021 Mar 14. PMID 33719603
- [Background] Pavana NAP, Ghosh AJEAB. Effectiveness of Core Stability Exercise and Proprioception Exercise on Balance in Subjects with Diabetic Neuropathy-A Randomized Controlled Trial. 2021;15(3):81.
- [Background] Jeon MJ, Jeon HS, Yi CH, Kwon OY, You SH, Park JH. Block and Random Practice: A Wii Fit Dynamic Balance Training in Older Adults. Res Q Exerc Sport. 2021 Sep;92(3):352-360. doi: 10.1080/02701367.2020.1733456. Epub 2020 May 13. PMID 32401683
- [Background] Cavalcante Neto JL, Steenbergen B, Wilson P, Zamuner AR, Tudella E. Is Wii-based motor training better than task-specific matched training for children with developmental coordination disorder? A randomized controlled trial. Disabil Rehabil. 2020 Sep;42(18):2611-2620. doi: 10.1080/09638288.2019.1572794. Epub 2019 Feb 22. PMID 30794762
- [Background] Kaur S, Koley SJJ. Effectiveness of trunk balance exercises and wii fit TM balance exercises in managing disability and pain in patients with chronic low back pain. 2019.
- [Background] Marques-Sule E, Arnal-Gomez A, Buitrago-Jimenez G, Suso-Marti L, Cuenca-Martinez F, Espi-Lopez GV. Effectiveness of Nintendo Wii and Physical Therapy in Functionality, Balance, and Daily Activities in Chronic Stroke Patients. J Am Med Dir Assoc. 2021 May;22(5):1073-1080. doi: 10.1016/j.jamda.2021.01.076. Epub 2021 Feb 24. PMID 33639116
- [Background] Cicek A, Ozdincler AR, Tarakci E. Interactive video game-based approaches improve mobility and mood in older adults: A nonrandomized, controlled tri̇al. J Bodyw Mov Ther. 2020 Jul;24(3):252-259. doi: 10.1016/j.jbmt.2020.01.005. Epub 2020 Feb 6. PMID 32825997
- [Background] Cimino V, Chisari CG, Raciti G, Russo A, Veca D, Zagari F, Calabro RS, Patti F. Objective evaluation of Nintendo Wii Fit Plus balance program training on postural stability in Multiple Sclerosis patients: a pilot study. Int J Rehabil Res. 2020 Sep;43(3):199-205. doi: 10.1097/MRR.0000000000000408. PMID 32371848
- [Background] Watkhuma A, Boonyaroma O, Srisupornkornkoolb K. Effect of Wii Balance Board and motor imagery on balance and muscle strength in football players
- [Background] Yuan RY, Chen SC, Peng CW, Lin YN, Chang YT, Lai CH. Effects of interactive video-game-based exercise on balance in older adults with mild-to-moderate Parkinson's disease. J Neuroeng Rehabil. 2020 Jul 13;17(1):91. doi: 10.1186/s12984-020-00725-y. PMID 32660512
- [Background] Hung ES, Chen SC, Chang FC, Shiao Y, Peng CW, Lai CH. Effects of Interactive Video Game-Based Exercise on Balance in Diabetic Patients with Peripheral Neuropathy: An Open-Level, Crossover Pilot Study. Evid Based Complement Alternat Med. 2019 Mar 6;2019:4540709. doi: 10.1155/2019/4540709. eCollection 2019. PMID 30956680
- [Derived] Rehman SSU, Hassan D, Ikram M, Ikram M. Effects of Wii Fit-based Exercises versus proprioceptive training on balance and fall risk in patients with diabetic neuropathy. Pak J Med Sci. 2025 Feb;41(2):393-398. doi: 10.12669/pjms.41.2.8775. PMID 39926688